CLINICAL TRIAL: NCT03134144
Title: Chairless Chair Exoskeleton. Work-physiological-biomechanical Analysis of the Lower Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Tessy Luger, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UKT-2017-AS0-1569
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: Exoskeleton; Manual materials handling; Musculoskeletal disorders; Posture; Standing work; Muscle activity
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First without exoskeleton then with exoskeleton (Experimental): Subject will perform the conditions as described under "model description" first without the exoskeleton and then with the exoskeleton.
  Interventions: Device: Exoskeleton "Chairless Chair"
- First with exoskeleton then without exoskeleton (Experimental): Subject will perform the conditions as described under "model description" first with the exoskeleton and then without the exoskeleton.
  Interventions: Device: Exoskeleton "Chairless Chair"

INTERVENTIONS:
Device: Exoskeleton "Chairless Chair" — One solution to reduce the exposure of employees to associated risks for developing work-related musculoskeletal disorders is to use exoskeletons. Using such a device in dynamic environments has the advantage over, e.g., robotics because it does not need any programming or teaching of robots. Moreover, exoskeletons are worn at the body and do not have to overcome spatial issues. In a recent review, 26 different exoskeletons have been described of which only two were designed to support the lower body during heavy work (de Looze et al. 2015). For lower intensive work tasks, like assembly tasks in the automobile industry, no study has focused on using exoskeletons to relieve employees while performing the work standing.

SUMMARY:
Standing work is associated with increased risks of venous and musculoskeletal disorders; particularly low back pain is commonly reported in prolonged standing work. In manufacturing work, workstations often do not allow standing aids due to insufficient functional and spatial conditions. In 2014, the car manufacturer Audi introduced the lower leg exoskeleton developed by Noonee to their employees working in the factories. This exoskeleton, the 'Chairless Chair' has the advantage that standing work can be performed while technically sitting on this device. The exoskeleton offers the potential for reduced awkward body postures, but it is unclear which physiological and biomechanical loads are influenced and how. This proposal provides a study design evaluating the 'Chairless Chair' in a laboratory setting, by testing its effectiveness in terms of physiological and biomechanical parameters. It is suggested to compare different assembly tasks while wearing the exoskeleton, compared with not wearing the exoskeleton. The 'Chairless Chair' is developed in one size only, which is why we propose to include participants of different body height, which will enable us to investigate whether body height influences the effectiveness of wearing the device.

DETAILED DESCRIPTION:
Each participant was exposed to all experimental conditions, which were the following:

* Standing without the exoskeleton
* Sitting with the exoskeleton

For both experimental conditions, the working height was adjusted to the individual to become optimal. The working distance to the simulated assembly tasks was also adjusted to the individual to become optimal. Both the working height and distance were based on textual guidelines provided in DIN EN ISO 14738:2009-07.

Each work cycle consisted of assembling and disassembling the following three tasks:

* Screwing
* Clip fitting
* Cable mounting

In addition, we investigated suboptimal working heights and distances. The results of these suboptimal conditions will not be reported in the results on this website, but in a separate publication.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 40 years old;
* Gender: male;
* Voluntary informed consent (oral and written) is obligatory for study participation.

Exclusion Criteria:

* Age: <18 and >40 years old;
* Gender: female;
* People under the influence of intoxicants, analgesics, or muscle relaxants;
* Alcohol abuse;
* People with cardiovascular diseases;
* People with a heart pacemaker;
* People with a disability who, due to their restriction at a workplace of this kind, will not be able to participate;
* People with Diabetes Mellitus;
* People with severe muscle contractions of the lower extremities, back or arms;
* People with acute ailments or pain;
* People who are unable to complete the examination program due to language or cognitive obstacles;
* Depending on the degree of severity, people with diseases of the veins and joints of the lower extremities, spine, muscle disorders, symptomatic neurological-psychiatric diseases, acute pain syndromes, maladies or other current diseases.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Occupational and Social Medicine and Health Services Research, University Hospital Tübingen, Faculty of Medicine, Eberhard Karls University Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Luger T, Seibt R, Cobb TJ, Rieger MA, Steinhilber B. Influence of a passive lower-limb exoskeleton during simulated industrial work tasks on physical load, upper body posture, postural control and discomfort. Appl Ergon. 2019 Oct;80:152-160. doi: 10.1016/j.apergo.2019.05.018. Epub 2019 May 30. PMID 31280799
- [Result] Luger T, Cobb TJ, Seibt R, Rieger MA, Steinhilber B. Subjective Evaluation of a Passive Lower-Limb Industrial Exoskeleton Used During simulated Assembly. IISE Transactions on Occupational Ergonomics and Human Factors, 2018.
- See also: Page 78: oral presentation of the study at the PREMUS 2019 conference in Bologna, Italy. — http://www.premus2019.com/wp-content/uploads/2019/09/PREMUS-2019-Abstact-30.08.19.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteering participants were recruited via the investigators that collaborated in this study.
Pre-assignment Details: None of the recruited volunteering participants was excluded based on the exclusion criteria.
  One subject dropped out prior to the measurement due to time constraints.
Groups:
- First Without Exoskeleton Then With Exoskeleton: Subject will perform the conditions as described under "model description" first with and then without the exoskeleton.
- First With Exoskeleton and Then Without Exoskeleton: Subject will perform the conditions as described under "model description" first with and then without the exoskeleton.
  Exoskeleton "Chairless Chair": One solution to reduce the exposure of employees to associated risks for developing work-related musculoskeletal disorders is to use exoskeletons. Using such a device in dynamic environments has the advantage over, e.g., robotics because it does not need any programming or teaching of robots. Moreover, exoskeletons are worn at the body and do not have to overcome spatial issues. In a recent review, 26 different exoskeletons have been described of which only two were designed to support the lower body during heavy work (de Looze et al. 2015). For lower intensive work tasks, like assembly tasks in the automobile industry, no study has focused on using exoskeletons to relieve employees while performing the work standing.
Period: Overall Study
Arm/Group | First Without Exoskeleton Then With Exoskeleton | First With Exoskeleton and Then Without Exoskeleton
Started | 15 | 30
Completed | 15 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Three additional subjects were recruited on top of the the sample size calculation, because three of the earlier measured subject had some missing data due to technical problems.
Groups:
- First Without Exoskeleton Then With Exoskeleton: Subject will perform the conditions as described under "model description" first without and then with the exoskeleton.
- First With Exoskeleton Then Without: Subject will perform the conditions as described under "model description" first with and then without the exoskeleton.
- Total: Total of all reporting groups
Arm/Group | First Without Exoskeleton Then With Exoskeleton | First With Exoskeleton Then Without | Total
Number analyzed (Participants) | 15 | 30 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (2.7) | 25.2 (3.0) | 24.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 30 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Center of Pressure
Description: Indicator for the balance of the study participants. This outcome was measured using a force plate, in which the anteroposterior and mediolateral directions of the center of pressure are recorded. The center of pressure is a visual projection of the center of mass of the participant. For the anteroposterior direction of the center of pressure, a positive value [mm] represents the anterior direction and a negative value [mm] represents the posterior direction. For the mediolateral direction of the center of pressure, a positive value [mm] represents the right-lateral direction and a negative value [mm] represents the left-lateral direction.
  For this outcome, we recorded the anteroposterior direction of the center of pressure.
  The outcome is in mm, where neg. reflects the posterior direction and pos. the anterior direction.
Time Frame: 10 minutes of 2 hours
Population: In total, two participants dropped out due to missing information with regard to the base of support, which is necessary to calculate the centre of pressure.
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- First With Exoskeleton and Then Without Exoskeleton: Subject will perform the conditions as described under "model description" first with the exoskeleton and then without the exoskeleton.
Arm/Group | First Without Exoskeleton Then With Exoskeleton | First With Exoskeleton and Then Without Exoskeleton
Number analyzed (Participants) | 14 | 29
mm
  Experimental conditions without exoskeleton | -42.76 [-48.19 to -25.55] | -34.98 [-49.16 to -22.18]
  Experimental conditions with exoskeleton | -118.34 [-128.42 to -107.43] | -122.16 [-130.80 to -111.58]

2. Primary Outcome: Muscle Activity of the Lower Back (M. Erector Spinae Lumbalis)
Description: Indicator for the muscular load in the lower back (M. erector spinae lumbalis) that may change when wearing the passive exoskeleton.
  The muscle activity was recorded using bipolar surface electromyography, during which two electrodes are placed on the muscle belly. The absolute value of muscle activity recordings is in microvolt, but since this is difficult to interpret, we have normalized this to a reference voluntary contraction that was executed by each participant prior to the experiment. The unit of measure for normalized muscle activity therefore is a percentage, i.e. a percentage of the electrical activity during the reference voluntary contraction [%RVE].
Time Frame: 10 minutes of 2 hours
Population: Data of 7 participants are missing due to failed data recordings.
Measure: Median (Inter-Quartile Range); unit: %RVE
Groups:
- First With Exoskeleton and Then Without the Exoskeleton: Subject will perform the conditions as described under "model description" first with the exoskeleton and then without the exoskeleton.
Arm/Group | First Without Exoskeleton Then With Exoskeleton | First With Exoskeleton and Then Without the Exoskeleton
Number analyzed (Participants) | 13 | 26
%RVE
  Experimental conditions without the exoskeleton | 11.02 [7.06 to 13.89] | 7.78 [6.62 to 11.70]
  Experimental conditions with the exoskeleton | 6.80 [5.39 to 11.11] | 8.29 [4.58 to 11.44]

3. Secondary Outcome: Back Posture: Upper Back Forward Flexion Angle With Respect to the Perpendicular (Earth)
Description: The posture of the back may indicate whether the relative body posture changed when wearing the passive exoskeleton compared to not wearing the passive exoskeleton.
  In the current study, back posture was recorded using two gravimetric position sensors placed on the thoracic vertebrae T3 and lumbal vertebrae L3.
  The difference between both position sensors represented the trunk forward flexion angle [°].
Time Frame: 10 minutes of 2 hours
Population: Data of 8 subjects is missing due to failed recordings.
Measure: Median (Inter-Quartile Range); unit: °
Arm/Group | First Without Exoskeleton Then With Exoskeleton | First With Exoskeleton Then Without Exoskeleton
Number analyzed (Participants) | 13 | 24
°
  Experimental conditions without the exoskeleton | 11.55 [4.83 to 17.10] | 5.10 [-3.31 to 10.83]
  Experimental conditions with the exoskeleton | 25.00 [14.89 to 36.85] | 20.95 [12.30 to 31.08]

4. Secondary Outcome: Subjective Feeling of Overall Discomfort
Description: Indicate whether participants develop feelings of discomfort in different experimental conditions when wearing or not wearing the passive exoskeleton.
  Discomfort was recorded using an 11-point numeric rating scale, running from 0 (no discomfort at all) to 10 (maximally imaginable discomfort).
  So, the outocme is in [units on a scale from 0 to 10].
Time Frame: 10 minutes of 2 hours
Population: All participants were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- First With Exoskeleton Then Without Exoskeleton: Subject will perform the conditions as described under "model description" with the exoskeleton.
  Exoskeleton "Chairless Chair": One solution to reduce the exposure of employees to associated risks for developing work-related musculoskeletal disorders is to use exoskeletons. Using such a device in dynamic environments has the advantage over, e.g., robotics because it does not need any programming or teaching of robots. Moreover, exoskeletons are worn at the body and do not have to overcome spatial issues. In a recent review, 26 different exoskeletons have been described of which only two were designed to support the lower body during heavy work (de Looze et al. 2015). For lower intensive work tasks, like assembly tasks in the automobile industry, no study has focused on using exoskeletons to relieve employees while performing the work standing.
Arm/Group | First Without Exoskeleton Then With Exoskeleton | First With Exoskeleton Then Without Exoskeleton
Number analyzed (Participants) | 15 | 30
units on a scale
  Experimental conditions without the exoskeleton | 0 [0 to 0] | 0 [0 to 1.25]
  Experimental conditions with the exoskeleton | 2 [0 to 2] | 0 [0 to 2]

5. Secondary Outcome: Participant Evaluation
Description: A questionnaire indicating whether wearing the passive exoskeleton during simluated assembly tasks is evaluated as comfortable, feasible, and usable.
  Below, the 10 statements questions as part of the participant evaluation questionnaire are shown with an interpretation of the score.
  1 generally reflects "I do not agree at all" whereas 10 generally reflects "I fully agree".
  Depending on the question, a score closer or equal to 1 is better and 10 worse, or vice versa.
  Statements 1-8: a higher score (i.e., close to 10) is considered better Statements 9-10: a lower score (i.e., close to 1) is considered better
Time Frame: 2 hours
Population: All participants could be included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | First Without Exoskeleton Then With Exoskeleton | First With Exoskeleton Then Without
Number analyzed (Participants) | 15 | 30
units on a scale
  The exoskeleton was comfortable | 6.4 (2.1) | 6.9 (1.9)
  The exoskeleton was easy to operate / handle | 8.4 (1.4) | 8.7 (1.3)
  I was able to work precisely with the exoskeleton | 9.1 (1.1) | 8.7 (1.3)
  The exoskeleton is suitable for the simulated task | 8.3 (1.8) | 8.1 (1.6)
  I can imagine working with the exoskeleton longer | 7.4 (2.2) | 6.9 (2.1)
  The working posture was comfortable in high sit | 5.9 (2.0) | 5.1 (2.0)
  The working posture was comfortable in low sit | 6.9 (2.2) | 7.2 (1.7)
  I felt safe to use the exoskeleton in high sit | 7.5 (2.1) | 6.6 (2.1)
  I felt safe to use the exoskeleton in low sit | 8.1 (1.9) | 7.8 (1.4)
  I wanted to change position in high sit | 6.3 (2.5) | 5.6 (2.9)
  I wanted to change position in low sit | 4.9 (2.6) | 5.0 (2.8)

ADVERSE EVENTS:
Time Frame: Through study completion, i.e. 1 day
Description: We performed a non-harmful experimental cross-over study. None of the subjects reported any adverse events.
Groups:
- Without Exoskeleton: Subject will perform the conditions as described under "model description" without the exoskeleton.
- With Exoskeleton: Subject will perform the conditions as described under "model description" with the exoskeleton.
Arm/Group | Without Exoskeleton | With Exoskeleton
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT03134144/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03134144/Prot_SAP_001.pdf